#### SUPER SHELF CONSENT FORM SAMPLE A

A multicomponent intervention in the hunger relief network to improve diet among adults experiencing food insecurity

I am here today from the University of Minnesota. You are invited to be in a research study on increasing the ease of choosing healthy foods at food shelves. You were selected as a possible participant because of your participation at this food shelf today. We ask that you read this form and ask any questions you may have before agreeing to be in the study.

### **BACKGROUND INFORMATION**

This study is being conducted by Dr. Caitlin E. Caspi, from the Department of Family Medicine and Community Health in the Medical School at the University of Minnesota Twin Cities Campus.

This study will look at whether making changes in the food pantry affects what foods clients choose. It will also look at whether clients experience changes in diet or cardiovascular disease risk over time.

If you agree to be in this study, we would ask you to do the following things:

- 1. Allow us to record the food you have selected from the food shelf today
- 2. Take a survey now, and again in one year.
- 3. Complete two dietary assessments over the phone in the next three weeks, and again in one year
- 4. Provide us with contact information so we can follow up with you to take the survey and two dietary assessments again.

The survey asks questions about you and your household, your visits to the food shelf, and your satisfaction with the food shelf. It also asks you to report your risk factors for cardiovascular disease (to the best of your knowledge). The survey takes about 10-15 minutes to complete. The dietary assessment asks you to list what you have eaten in the last 24 hours. It takes about 20-30 minutes and will be completed over the phone.

### RISKS AND BENEFITS OF BEING IN THE STUDY

<u>The study has minimal risk</u>; however, you may feel uncomfortable answering some of the questions on the survey. You do not have to answer a question if you do not want to. You will be able to take the survey in a private area. If for any reason you would like assistance taking the survey, a researcher can either give assistance or give the whole survey to you verbally in a private room.

We will keep your data locked and secured. Although it is unlikely, there is a possibility a data breach could occur and your data could be shared with those outside of the study team.

<u>There are no direct benefits</u> to you for participating in the study today. However, we are working towards making healthy foods more available and healthier food choices easier for food shelf clients.

#### **COMPENSATION**

For your participation in this study you will be given a Prepaid Debit card called ClinCard. Your card will be loaded as you complete study activities. You can receive up to \$45 now and an

IRB Code # Version Date: 12.29.17

Approved for used UMN IRB Effective on 2/15/2019 IRB Study Number: 1612S02201 additional \$45 in one year. We say "up to" because you will get different amounts based on which study tasks you complete.

# **COMPENSATION (CONTINUED)**

Today you can get:

• \$15 for completing a survey and shopping bag check

Within about three weeks you can get:

- \$15 for completing the first dietary assessment (within the next 10 days over the phone).
- \$15 for completing the second dietary assessment (over the phone within the next 20 days).

In one year we will contact you for 2 additional dietary assessments and a survey (up to \$45), which will be emailed to you.

- \$15 for the online survey
- \$15 for the first dietary assessment
- \$15 for the second dietary assessment

## **CONFIDENTIALITY**

The records of this study will be kept private. In any sort of report we might publish, we will not include any information that will make it possible to identify a subject. Research records will be stored securely and only researchers will have access to the records. Study data will be encrypted according to current University policy for protection of confidentiality.

### **VOLUNTARY NATURE OF THE STUDY**

Participation in this study is voluntary. Your decision whether or not to participate will not affect your current or future relations with the University of Minnesota or with the food shelf. If you decide to participate, you are free to not answer any question or withdraw at any time without affecting those relationships.

## **CONTACTS AND QUESTIONS**

You may ask any questions you have now. If you have questions later, **you are encouraged** to contact us:

- Principal Investigator, Dr. Caitlin Caspi at 612-626-7074 or cecaspi@umn.edu
- Project Manager, Kate Grannon, at 612-625-7179 youn1286@umn.edu or

If you have any questions or concerns regarding this study and would like to talk to someone other than the researcher(s), **you are encouraged** to contact the Research Participants' Advocate Line at 612-625-1650 or go to https://research.umn.edu/units/hrpp/research-participants/questions-concerns.

You will be given a copy of this information to keep for your records.

# STATEMENT OF CONSENT

I have read the above information. I have asked questions and have received answers. I consent to participate in the study.

IRB Code # Version Date: 12.29.17

Approved for used UMN IRB Effective on 2/15/2019 IRB Study Number: 1612S02201

| Signature: | Date: |
|------------|-------|
| Signature. | Datc. |